CLINICAL TRIAL: NCT06439459
Title: Quantitative Measurements of the Skin Dermal Regeneration After Stromal Vascular Fraction Transplantation
Brief Title: Skin Dermal Regeneration After Stromal Vascular Fraction Transplantation
Acronym: SDR-SVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shanghai9th-SDR-SVF-ZT; 22MC1940300 (Other Grant/Funding Number: Science and Technology Commission of Shanghai Municipality); shslczdzk00901 (Other Grant/Funding Number: Shanghai Municipal Key Clinical Specialty)
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2023-01

CONDITIONS: Skin Regeneration
Keywords: skin expansion; stromal vascular fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stromal vascular fraction transplantation (Experimental): Subcutaneous fat was harvested from either the abdomen or the posterior inner thigh region and then digested with 600 U of collagenase (Shanghai Qiaoyuan Biological Pharmaceutical Co., Ltd, Shanghai, China) at 37°C and 150rpm for three hours. After enzymatic digestion, the lower aqueous phase liquid was aspirated to acquire the stromal vascular fraction (SVF). The SVF cell-pellet was washed and adjusted to 2×10^6 cells/mL. The skin was marked with methylene blue and a total of 0.5ml (around 1×10^6 cells) were transplanted intradermally at the center of each 2cm×2cm squares.
  The expander was inflated two times a week using constant pressure inflation method, where the intracapsular pressure was monitored using a pressure meter and the inflation was halted when the pressure reached 100 mmHg. This procedure was repeated until adequate skin area was achieved for subsequent facial restoration surgery.
  Interventions: Procedure: Stromal vascular fraction transplantation

INTERVENTIONS:
Procedure: Stromal vascular fraction transplantation — Stromal vascular fraction was extracted from subcutaneous fat harvested from either the abdomen or the posterior inner thigh region. The SVF cell-pellet was washed and was adjusted to 2×10^6 cells/mL. The skin was marked with methylene blue and a total of 0.5ml (around 1×10^6 cells) were transplanted intradermally at the center of each 2cm×2cm squares.
  The expander was inflated two times a week using constant pressure inflation method, where the intracapsular pressure was monitored using a pressure meter and the inflation was halted when the pressure reached 100 mmHg. This procedure was repeated until adequate skin area was achieved for subsequent facial restoration surgery.

SUMMARY:
This study is a prospective, exploratory investigation aimed at exploring the efficacy of stromal vascular fraction (SVF) transplantation in treating exhaustion of dermal regenerative capacity during skin expansion. The dermal thickness, texture, and perfusion before and after SVF transplantation would be recorded and analyzed by a series of quantitative devices including laser 3D scanner, Doppler ultrasound, VISIA skin analyzer, CK skin analyzer, and indocyanine green angiography.

DETAILED DESCRIPTION:
This study is a prospective, exploratory investigation aimed at exploring the efficacy of stromal vascular fraction (SVF) transplantation in treating exhaustion of dermal regenerative capacity during skin expansion. The dermal thickness, texture, and perfusion before and after SVF transplantation would be recorded and analyzed by a series of quantitative devices including laser 3D scanner, Doppler ultrasound, VISIA skin analyzer, CK skin analyzer, and indocyanine green angiography.

The trial aims to include patients experiencing dermal exhaustion during the process of skin soft tissue expansion. We will extract SVF components from autologous adipose tissue and injected intradermally into the expanded skin. The changes of dermis of expanded skin were recorded before the treatment (baseline), and at 4 weeks and 8 weeks follow-up timepoints after SVF transplantation. More specifically, skin surface area was measured using laser 3D scan; skin thickness and texture were detected by Doppler ultrasound, VISIA skin analyzer and CK skin analyzer; skin blood perfusion was analyzed using indocyanine green angiography.

ELIGIBILITY:
Inclusion Criteria:

* had undergone tissue expansion treatment;
* show signs of deterioration of skin texture during expansion, including stretch marks or thinning of the dermis (<2mm) with no improvement after suspending expansion for 2 weeks;
* require further expansion to achieve the size for defect reconstruction.

Exclusion Criteria:

* Patients with serious underlying diseases such as cardiovascular or cerebrovascular disease, peripheral vascular disease, or impaired liver or kidney function;
* Patients with a long history of smoking and alcohol use who have not quit smoking or drinking;
* Patients allergic to iodine or iodine-containing preparations;
* Patients with psychiatric disorders, lack of insight, or those who cannot accurately express themselves or cooperate;
* Patients with contraindications for SVF transplantation, such as ulceration or infection of the expanded skin;
* Patients with severely loose skin or insufficient subcutaneous fat tissue;
* Patients who request to withdraw informed consent and exit the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Dermal thickness | Baseline: before SVF transplantation (Baseline); Follow-up: 4 and 8 weeks after SVF transplantation
  Using Doppler ultrasound to measure the full-thickness of skin dermis of the expanded skin. The measurements were conducted at the center of the expanded skin and other four points (above, below, left, right) around the center. The average value is taken to represent the dermal thickness of the patient's expanded skin.

SECONDARY OUTCOMES:
Skin surface area | Baseline: before SVF transplantation (Baseline); Follow-up: 4 and 8 weeks after SVF transplantation
  Using the HSCAN771 handheld laser 3D scanner and the VIVID910 3D laser scanning system to measure the surface area of the expanded skin.

OTHER OUTCOMES:
Skin texture (dermal rupture) | Baseline: before SVF transplantation (Baseline); Follow-up: 4 and 8 weeks after SVF transplantation
  Using the VISIA skin analyzer to visualize the distribution of dermal marks, which is an indication of dermal rupture. Briefly, photographs of the patient's expanded skin were taken from three standard angles: front, left side, and right side. Use the VISIA instrument to generate texture imaging of the expanded skin, selecting the expanded skin and surrounding normal skin as the region of interest. Employ the instrument's built-in red area analysis function to analyze the distribution of dermal marks in the expanded skin.
Skin texture (elasticity) | Baseline: before SVF transplantation (Baseline); Follow-up: 4 and 8 weeks after SVF transplantation
  Using the elasticity probe (Cutometer® MPA 580) of CK Skin analyzer to measure the elasticity of the expanded skin. Represent skin softness through the skin viscoelasticity parameter R2 (R2 = Ua/Uf, where Ua is the total elastic and plastic recovery, and Uf is the total elastic and plastic deformation). An R2 value closer to 1 indicates better skin elasticity. The measurements were conducted at the center of the expanded skin and other four points (above, below, left, right) around the center. Each point is measured three times, and the average value is taken to represent the measurement for that point.
Skin perfusion | Baseline: before SVF transplantation (Baseline); Follow-up: 4 and 8 weeks after SVF transplantation
  Indocyanine green (ICG) angiography was used to detect the blood perfusion of the expanded skin. Briefly, the detector of SPY imaging system was adjusted to approximately 20 cm from the surface of the flap. A white light photograph of the expanded skin was taken. Without changing the detector position, indocyanine green imaging was performed as follows: Inject 2 ml of ICG solution (2.5 mg/ml) intravenously and fluorescence signals from the expanded skin were collected by SPY imaging system. The integrated SPY-Q software was used for the analysis of the arterial and venous perfusion of the expanded flap.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Huangpu, China

IPD SHARING:
Plan to Share IPD: No
Any additional information regarding individual participants is available from the principle investigator of this study upon reasonable request.